CLINICAL TRIAL: NCT04822961
Title: A Randomized, Double-Blinded, Placebo-Controlled, Multicenter, Phase II Study to Evaluate Senaparib in mCRPC Patients With Homologous Recombination Repair Gene Alterations After Docetaxel Treatment
Brief Title: Senaparib in mCRPC Patients With Homologous Recombination Repair Gene Alterations After Docetaxel Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Impact Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMP4297-202
Record Dates: First submitted 2020-09-03; First posted 2021-03-30 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: mCRPC
MeSH Terms: interventions — senaparib

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blinded, Placebo-Controlled
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Senaparib (IMP4297) 20 mg (Experimental): During the treatment period, eligible patients will receive single agent of Senaparib at a dose of 100 mg once daily (QD), continuously on a 4-week cycle
  Interventions: Drug: Placebo
- Placebo (Placebo Comparator): During the treatment period, eligible patients will receive placebo QD, continuously on a 4-week cycle
  Interventions: Drug: Senaparib

INTERVENTIONS:
Drug: Placebo — Senaparib-matched placebo capsules
  Arms: Senaparib (IMP4297) 20 mg
Drug: Senaparib — 20 mg capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Senaparib in metastatic castration-resistant prostate cancer (mCRPC) patients with homologous recombination repair (HRR) gene alterations after docetaxel treatment

DETAILED DESCRIPTION:
This is a randomized, double-blinded, placebo-controlled, multicenter, Phase II study in mCRPC patients with HRR gene alterations after docetaxel therapy to evaluate the anti-tumor activity and safety of Senaparib.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must voluntarily participate in this clinical study. Be willing written informed consent form (ICF) prior to any study activity.
2. Male ≥18 years of age on the day of signing the ICF.
3. Patients must have histologically or cytologically confirmed prostate adenocarcinoma.
4. Surgically or medically castrated, with serum testosterone levels of ≤50 ng/dL (≤1.73 nmol/L). If the patient is being treated with LHRH agonists/antagonists (patient who have not undergone orchiectomy), this therapy must be continued throughout the study.
5. Patients have adequate organ functions, as indicated by the following laboratory values (had not received blood transfusion, apheresis infusion, erythropoietin, granulocyte colony-stimulating factor (G-CSF), and other relevant medical support within 14 days before the administration of study drug).
6. Patients have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
7. Male patients must use a condom during treatment and for 3 months after the last dose of study drug when having sexual intercourse with a woman of childbearing potential. Female partners of male patients should also use an acceptable method of contraception if they are of childbearing potential.

Exclusion Criteria:

1. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
2. Prior treatment with a polyadenosine 5'diphosphoribose polymerisation (PARP) inhibitor, including Senaparib.
3. Patients with a known hypersensitivity to Senaparib or any of the component of Senaparib.
4. Initiating bisphosphonate/denosumab therapy or adjusting bisphosphonate/denosumab dose/regimen within 28 days prior to the first dose of study drug. Patients on a stable bisphosphonate/denosumab regimen are eligible and may continue.
5. Patients who have received strong inhibitors/inducers of CYP3A4 which cannot be discontinued 21 days prior to the first dose of study drug and withheld throughout the study drug treatment. Patients received phenobarbital/enzalutamide will require a 5-week washout prior to the first dose of study drug.
6. Patients with MDS or AML, or with clinical features suggestive of MDS or AML.
7. Patients with serious acute or chronic infections.
8. Patients who have received a live virus or bacterial or RNA vaccination within 28 days prior to the first dose of study drug.
9. Patients are unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Estimated)
Dates: Start 2021-12-31 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
rPFS assessed by BICR | 80 weeks
  To evaluate the impact of Senaparib on radiographic progression free survival (rPFS), compared with the placebo, in metastatic castration-resistant prostate cancer (mCRPC) patients with BRCA1/2 gene alteration who have not progressed after docetaxel therapy assessed by Blinded Independent Central Review (BICR).

SECONDARY OUTCOMES:
rPFS assessed by BICR | 80 weeks
  To evaluate the impact of Senaparib on rPFS, compared with the placebo, in mCRPC patients with homologous recombination repair (HRR) gene alterations who have not progressed after docetaxel therapy assessed by BICR.
Time to pain progression | 80 weeks
  To evaluate the impact of Senaparib on time to pain progression, compared with the placebo, in mCRPC patients with BRCA1/2 gene alteration who have not progressed after docetaxel therapy.
Time from randomization to the first SSRE | 80 weeks
  To evaluate the impact of Senaparib on time to the first symptomatic skeletal related events (SSRE), compared with the placebo, in mCRPC patients with BRCA1/2 gene alteration who have not progressed after docetaxel therapy.
OS | 80 weeks
  To evaluate the impact of Senaparib on overall survival (OS), compared with the placebo, in mCRPC patients with BRCA1/2 gene alteration who have not progressed after docetaxel therapy.
PFS2 | 80 weeks
  To evaluate the impact of Senaparib on second progression (PFS2), compared with the placebo, in mCRPC patients with BRCA1/2 gene alteration and HRR gene alterations who have not progressed after docetaxel therapy.
Time to pain progression | 80 weeks
  To evaluate the impact of Senaparib on time to pain progression, compared with the placebo, in mCRPC patients with HRR gene alterations who have not progressed after docetaxel therapy.
Time from randomization to the first SSRE | 80 weeks
  To evaluate the impact of Senaparib on time to the first SSRE, compared with the placebo, in mCRPC patients with HRR gene alterations who have not progressed after docetaxel therapy.
OS | 80 weeks
  To evaluate the impact of Senaparib on OS, compared with the placebo, in mCRPC patients with HRR gene alterations who have not progressed after docetaxel therapy.
rPFS assessed by the investigator | 80 weeks
  To evaluate the impact of Senaparib on rPFS assessed by the investigator, compared with the placebo, in mCRPC patients with BRCA1/2 gene alteration and HRR gene alterations who have not progressed after docetaxel therapy.
Time to PSA progression | 80 weeks
  To evaluate the impact of Senaparib on time to prostate-specific antigen (PSA) progression, compared with the placebo, in mCRPC patients with BRCA1/2 gene alteration and HRR gene alterations who have not progressed after docetaxel therapy.
Objective response rate (ORR) according to RECIST v1.1 assessed by BICR | 80 weeks
  To evaluate the impact of Senaparib on radiographic response rate assessed by BICR, compared with the placebo, in mCRPC patients with BRCA1/2 gene alteration and HRR gene alterations who have measurable lesion and have not progressed after docetaxel therapy.
Objective response rate (ORR) according to RECIST v1.1 assessed by investigator | 80 weeks
  To evaluate the impact of Senaparib on radiographic response rate assessed by the investigator, compared with the placebo, in mCRPC patients with BRCA1/2 gene alteration and HRR gene alterations who have measurable lesion and have not progressed after docetaxel therapy.
PSA response rate according to PCWG3 criteria assessed by central laboratory | 80 weeks
  To evaluate the impact of Senaparib on PSA response rate, compared with the placebo, in mCRPC patients with BRCA1/2 gene alteration and HRR gene alterations who have not progressed after docetaxel therapy.
Safety endpoints | 80 weeks
  Number of participants with treatment-related adverse events as assessed by NCI CTCAE v5.0.
Cmax | 80 weeks
  Maximum plasma concentration，To characterize the plasma PK profile of Senaparib via population PK (popPK) modeling

CONTACTS AND LOCATIONS:
Locations (6):
- Our lady of Lourdes Urology, Binghamton, New York, United States
- Australia (4):
  - Princess Alexandra Hospital, Brisbane
  - Cabrini Hospital, Melbourne
  - Macquarie University Hospital, Sydney
  - John Flynn Hospital, Tugun
- IMPACT Therapeutics Inc., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No